CLINICAL TRIAL: NCT06404138
Title: Recovery From Disability After Geriatric-home Rehabilitation Versus Standard of Care: Pilot Study for a Randomised Multicentre Parallel Group Pragmatic Trial in Older Persons With Disability at Hospital Discharge.
Brief Title: Recovery From Disability After Geriatric-home Rehabilitation Versus Standard of Care: Pilot Study
Acronym: RECOVER@HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: CHU UCL Namur (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S65872; KCE22-1383 (Other Grant/Funding Number: KCE)
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Disability Physical
Keywords: Disability; Geriatric; Rehabilitation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients are randomized 1:1 in one of the two intervention groups
Who Masked: Outcomes Assessor
Masking Description: The study nurse, who assesses the outcomes during home visits (baseline, after six weeks, after one year) will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receives 18 physiotherapy sessions at home over 6 weeks according to the Geriatric Activation program Pellenberg (GAPP, see intervention)
  Interventions: Other: The Geriatric Activation Program (GAPP) Home version
- Control group (Other): Older persons in the control group receive the standard of care, without any restrictions. This implies that some of the older persons in the control group could receive physical therapy, but the standard of care implies that although geriatricians regularly prescribe physical therapy the therapy is actually not started in most cases. Therefore, physical therapy will not often be delivered in the control group, and if it is delivered it will be less structured and at lower intensity and/or frequency. Moreover, physical therapy delivered to participants in the control group will not be supported by a targeted rehabilitation plan and a specific training for the therapists.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: The Geriatric Activation Program (GAPP) Home version — The rehabilitation at home intervention consists of three 45 minutes session per week (total of 18 sessions) with a different focus for each session. The therapy is goal-oriented and includes functional exercises in the home where possible (e.g. transfers such as getting out of bed, walking to the toilet etc.). There are three sessions per week: 1 for training strength, 1 for training balance and 1 for speed, coordination and endurance. Each session will start with gait rehabilitation as a warming-up.
  For each session, a set of exercises with varying levels of difficulty is available. As rehabilitation needs are diverse, the therapist is expected to choose the most appropriate exercise and the difficulty level of the exercise for the individual older person. This also includes scaling the exercises to the individual progression of the older person.
  Arms: Intervention group
Other: Standard of care — Standard of care, without any restrictions.
  Arms: Control group

SUMMARY:
At discharge after a hospitalization, many older people are not as able as before their hospital stay and have difficulty performing their daily activities at home. For example, washing and dressing themselves, housework or shopping are often more difficult after discharge from hospital. However, most older people do not receive any support in regaining their physical status and self-reliance. As a result, they often need permanent help from informal or professional caregivers. Their quality of life is also impacted and they have an increased risk of new hospital admissions.

Rehabilitation centers and hospital rehabilitation wards help the elderly to regain their daily functioning, but the number of places is very limited. This means that support for home rehabilitation is necessary for the vast majority of older people (almost 82,000 people per year). However, most of the time there is no support for home rehabilitation and the effect of such home rehabilitation programs has been little studied. Although studies show that home rehabilitation can improve physical functioning, the effect on impairments in daily activities and the quality of life of older people are not clear.

In a future multicenter RCT, the investigators want to study whether training and guidance by a physiotherapist contributes to the recovery of older people after discharge from hospital.

Patients will either receive standard care after hospitalization discharge, or intensive guidance from a physiotherapist. The patients guided by the physiotherapist are trained and supervised three times a week, for six weeks, to improve their muscle strength, balance, walking and mobility. The aim of the intensive home rehabilitation program is that the individual benefits from it in the longer term. Therefore, whether individuals who received the program are less limited in their daily functioning than those who did not receive the intensive rehabilitation program is checked after six months. In addition, the quality of life, physical functioning and healthcare costs for these two groups are also compared.

To ensure that the study is feasible, a small pilot study will first be performed. Here, the aim is to assess the feasibility of recruitment (screening and retaining participants, reasons for refusal and participant profiles), study procedures and intervention. This includes time registration by the study team and physiotherapists, assessment of study burden and experiences with the execution of the protocol. The findings of this pilot study will help deciding about progressing to a future definitive RCT.

ELIGIBILITY:
Inclusion Criteria:

* 75 years of age or older;
* disability (i.e., dependent in one or more activities of daily living) at hospital discharge;
* rehabilitation potential;
* capable of giving informed consent, and also giving their consent;

Exclusion Criteria:

* discharged to a nursing home or rehabilitation centre;
* receiving palliative care;
* enrolled in a specialised rehabilitation programme, e.g. cardiac rehabilitation, stroke rehabilitation, respiratory rehabilitation for COPD, and oncology rehabilitation;
* in active follow-up with a physical therapist, and for whom participation in the intervention would be too demanding or would compromise the integrity of the therapy and its anticipated outcomes.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment - screening | 1 year
  The number of potential participants screened/not screened for inclusion.
Feasibility of recruitment - retainment | 1 year
  The number of (potential) participants recruited/not recruited, randomised and retained (frequency and proportion of participants that are randomized and completed 6w follow up).
Feasibility of recruitment - reasons for non-participation | 1 year
  Potential participants' reasons for refusing to participate (qualitative), expressed in frequency per reason for declining participation.
Feasibility of study procedures, assessments and data collection | 1 year
  Assessment will focus on the timeliness and practicality of the randomisation, assessment and the data collection in the participants' home, processing and managing the data and study administration. This endpoint is assessed through interviewing study staff about their experiences.
Study participants' experience with the intervention | 1 year
  Semi-structured interviews with participants, assessing how the intervention did or did not meet their needs, intervention elements they did or did not appreciate, their perceived adherence to the therapy sessions, the level of difficulty of intervention elements in relation to their level of disability, the support from their therapist, the perceived benefit or lack thereof, their reasons for engaging or discontinuing the intervention, and reasons for (not) recommending the intervention to others in the same position.
Physical therapists' experience with the intervention | 1 year
  Interviews with physical therapists, addressing feasibility with a view to alternative elements of the intervention, the target group, the setting and their professional capabilities and limitations. Questions will also explore their experience with the adherence of the participants, and their perceptions regarding factors that influenced this.

SECONDARY OUTCOMES:
The profiles of study participants | 1 year
  Demographic information
Time spent on study procedures and assessments | 1 year
  The study nurses and medical doctors participating in the study will log the time they spend on the study in an electronic logbook. This will be done for patient 5 to 12 at each site. Time will be recorded in minutes per day, and will be stratified for screening, informed consent, randomisation, baseline visit, visit at 6 weeks follow-up, administration, and other. Data will be gathered up to six weeks when the intervention protocol is completed and follow-up data at six weeks are gathered. The endpoint will be expressed as the median time to complete the study procedures per participant.
The study burden for participants (older persons) | 6 weeks
  Audio recorded interviews using open-ended questions will focus on understanding how persons experience study participation and which aspects of the study might be perceived as hindrances or barriers in relation to their daily lives.Second, a modified version of the Perceived Research Burden Assessment instrument (5-point Likert scales) is used to quantify the study burden for individual participants.
The study burden for healthcare professionals | 1 year
  Structured interviews, focusing on understanding how they experienced screening for eligibility and how this could be disruptive for their daily practice.
Physical therapists' experiences with the training protocol | 1 year
  Physical therapists' experiences with the training needed to deliver the rehabilitation protocol will be assessed in a structured interview. Interview questions will focus on the format, the delivery, the content, and the duration of the training. Participants will also be asked to suggest changes or improvements. The interview is performed online and after completion of the training, and is audio recorded.
Blinding of outcome assessors | 1 year
  Structured interview addressing for which participants the study nurses feel they know, suspect or do not know to which group a person was randomized, and -if relevant- how they found out. Nurses' ideas of group allocation will be checked against the actual group allocation. This information will be used to construct a Blinding Index. This endpoint will be expressed as the frequency and proportion of participants where blinding was not achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Theo van Achterberg, MSc, PhD, Principal Investigator — KU Leuven
Locations (2):
- Belgium (2):
  - CHU UCL Namur, Godinne
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No
IPD will be shared upon publication of the primary endpoint of the full trial, which will have a separate registration on clinicaltrial.gov.

REFERENCES:
- [Derived] Van Grootven B, van Dijk M, Islam F, Coucke B, Fieuws S, Van Pottelbergh G, Flamaing J, Van Den Noortgate N, Velghe A, De Cock AM, Gillain S, Meeuwissen J, Bautmans I, Beckwee D, de Saint-Hubert M, van Uffelen J, Schoevaerdts D, Tournoy J, van Achterberg T. Recovery from disability after geriatric-home rehabilitation versus standard of care: protocol for a pilot study in older persons with disability at hospital discharge. Pilot Feasibility Stud. 2025 Jun 21;11(1):87. doi: 10.1186/s40814-025-01668-8. PMID 40544287
- See also: Trial description on funder web page — https://kce.fgov.be/en/recoverhome-recovery-from-disability-after-geriatric-home-rehabilitation-versus-standard-of-care-a